CLINICAL TRIAL: NCT06784206
Title: An Exploratory Clinical Study of Adebrelimab Maintenance Treatment Following Concurrent Chemoradiotherapy with Hyperfractionated Radiotherapy in Patients with Limited-Stage Small Cell Lung Cancer
Brief Title: Adebrelimab Maintenance Therapy After Concurrent Chemoradiotherapy with Hyperfractionated Radiotherapy in Limited-Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Anhui Shi, MD, Chief Physician, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024YJZ163
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Small Cell Lung Cancer, Limited Stage; Hyperfractionated Accelerated Radiotherapy; Simultaneous Radiotherapy and Chemotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): In this study, patients will receive concurrent hyperfractionated accelerated radiotherapy (HART) combined with chemotherapy for 4 cycles. If patients achieve a complete response (CR) or partial response (PR) after the initial treatment, they will be given prophylactic cranial irradiation (PCI). Following PCI, patients will enter the maintenance treatment phase with Adebrelimab, which will continue until disease progression, death, or the development of intolerable toxicity.
  Interventions: Drug: Adebrelimab Maintenance Therapy After Concurrent Chemoradiotherapy with Hyperfractionated Radiotherapy

INTERVENTIONS:
Drug: Adebrelimab Maintenance Therapy After Concurrent Chemoradiotherapy with Hyperfractionated Radiotherapy — Chemotherapy:
  Etoposide will be administered intravenously at a dose of 100 mg/m² on days 1 to 3 of each cycle. Cisplatin will be given at a dose of 75 mg/m² on day 1 of each cycle. The treatment will be repeated every 3 weeks for a total of 4 cycles.
  Concurrent Radiotherapy:
  Chest radiotherapy will be initiated concurrently with the first 3 cycles of chemotherapy. The total dose of radiotherapy will be 54 Gy, delivered in 30 fractions, with 2 fractions per day.
  Prophylactic Cranial Irradiation (PCI):
  For patients who achieve a partial response (PR) or complete response (CR) after chemoradiotherapy, PCI will be administered 3 to 4 weeks after the completion of chemoradiotherapy. The dose for PCI will be 25 Gy in 10 fractions.
  Adebrelimab Maintenance Therapy:
  Following PCI, patients will receive maintenance therapy with Adebrelimab. The dose will be 1200 mg administered intravenously on day 1 of each cycle. The treatment will be repeated every 3 weeks until disease progression, death

SUMMARY:
Small cell lung cancer (SCLC) remains a challenging disease with poor prognosis and limited treatment options despite decades of research. SCLC is an immunogenic tumor, and the use of T-cell immune checkpoint inhibitors targeting the PD-1/PD-L1 axis has shown promising antitumor activity, potentially extending patient survival. The combination of concurrent chemoradiotherapy followed by immune maintenance therapy has demonstrated significant efficacy in limited-stage SCLC. Moreover, hyperfractionated accelerated radiotherapy (HART) has been shown to improve overall survival in limited-stage SCLC compared to standard dose radiotherapy without increasing toxicity. However, there is a lack of exploration into the use of immune checkpoint inhibitors following concurrent chemoradiotherapy with HART in limited-stage SCLC.

This exploratory clinical study aims to investigate the efficacy and safety of adebrelimab maintenance treatment following concurrent chemoradiotherapy with HART in patients with limited-stage SCLC through a single-arm, open-label, prospective, single-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years, both genders are eligible;
* Histologically or cytologically confirmed limited-stage small cell lung cancer (according to the 8th edition of AJCC staging);
* Patients who have previously received no more than 2 cycles of standard chemotherapy or are treatment-naive;
* ECOG performance status: 0-1;
* Presence of measurable lesions according to RECIST 1.1 criteria (for RECIST 1.1 criteria, the longest diameter of tumor lesions on CT scan ≥10mm, and the shortest diameter of lymph node lesions on CT scan ≥15mm);
* Estimated life expectancy of at least three months;
* Participants must have adequate pulmonary function;

Normal function of major organs, which means meeting the following criteria:

Complete blood count:

Hemoglobin (HGB) ≥90 g/L; Absolute neutrophil count (ANC) ≥1.5×10⁹/L; Platelet count (PLT) ≥100×10⁹/L; White blood cell count (WBC) ≥3.0×10⁹/L;

Biochemical tests:

Serum albumin (ALB) ≥30 g/L; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3×ULN; Total bilirubin (TBIL) ≤1.5×ULN; this does not apply to patients diagnosed with Gilbert's syndrome (persistent or recurrent hyperbilirubinemia [mainly unconjugated bilirubin], without evidence of hemolysis or liver pathology). After consultation with a physician, patients with this condition may be allowed to participate in the study.

* Creatinine ≤1.5×ULN;
* Women of childbearing potential must have taken reliable contraceptive measures or have had a negative pregnancy test (serum or urine) within 7 days before enrollment. Both men and women of childbearing age must agree to take adequate contraceptive measures throughout the study period and for 6 months after the end of treatment;
* Participants voluntarily join this study, sign the informed consent form, have good compliance, and cooperate with follow-ups.

Exclusion Criteria:

* Histological mixture of SCLC and NSCLC components;
* Extensive-stage SCLC;
* Patients with a history of allogeneic organ transplant or allogeneic hematopoietic stem cell transplant or planned for transplant;
* Use of immunosuppressive drugs (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor drugs) within 14 days before the first use of Adebrelimab, excluding nasal and inhaled corticosteroids or physiologic doses of systemic corticosteroids (i.e., no more than 10 mg/day of prednisolone or equivalent physiologic dose of other corticosteroids);
* Known allergy to etoposide, cisplatin, Adebrelimab, or drug excipients; or severe allergic reactions to other monoclonal antibodies; Vaccination with live attenuated vaccines within 4 weeks before the first dose or planned during the study period;
* Presence of any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism) is not eligible. Exceptions to this criterion include:

Patients with vitiligo or alopecia;

* Patients with stable hypothyroidism under hormone replacement therapy (e.g., after Hashimoto's syndrome);
* Participants undergoing systemic treatment with bronchodilators, with unsatisfactory asthma control, are not eligible (those who had complete remission of asthma in childhood and require no intervention in adulthood may be included);
* Urinalysis showing proteinuria ≥++, or confirmed 24-hour urine protein ≥1.0g;

Previously diagnosed with any other malignancy, except for the following conditions:

* Adequately treated basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix;
* Malignancies treated with curative intent, with no known active disease for ≥5 years before the first dose in the study and with a low potential risk of recurrence;
* Infection with human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS);
* Within 6 months before enrollment, occurrence of the following conditions: myocardial infarction, severe/unstable angina, NYHA class 2 or higher heart failure, poorly controlled arrhythmias (including QTcF interval >450 ms for males, >470 ms for females, QTcF interval calculated by Fridericia formula), symptomatic congestive heart failure;
* Infections requiring drug intervention (e.g., intravenous antibiotics, antifungal, or antiviral drugs) within 4 weeks before the first dose, or unexplained fever ≥38.5°C during the screening period or before the first dose;
* Active tuberculosis, hepatitis B (HBV-DNA ≥500 IU/ml), hepatitis C (positive hepatitis C antibody, and HCV-RNA above the lower limit of detection of the analytical method), or co-infection with hepatitis B and C;
* Participation in any other drug clinical trial within 4 weeks before the first dose; Known history of abuse of psychoactive drugs or drug addiction;
* Presence of other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participation in the study, interfere with the study results, or patients whom the investigator deems unsuitable for participation in this study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events | Duration of treatment and follow up until death or 90 days after enrollment
  Treatment-related adverse events according to CTCAE 5.0

SECONDARY OUTCOMES:
PFS | From enrollment to the end of treatment at 1 and 2 year
  From the date of enrollment to the date of disease progression
OS | From date of enrollment to maximum of 2 years or death
  from the date of enrollment until death by any cause or last follow-up
ORR | From date of enrollment to maximum of 2 years
  The proportion of subjects with Best Overall Response (BOR) assessed as Complete Response (CR) or Partial Response (PR) according to RECIST 1.1 criteria
DCR | From date of enrollment to maximum of 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease (SD) based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes